CLINICAL TRIAL: NCT01987934
Title: Comparison of Morphometric Assessment Using Methyl Green Pyronin and AgNOR Staining of Oral Squamous Cell Carcinoma
Acronym: OSCC
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Academy of Interdisciplinary Dental Education and Research (Other)
Collaborators: Postgraduate Medical Institute, Lahore (Other)
Responsible Party: Principal Investigator, Ali Raza, Dr. Ali Raza, Academy of Interdisciplinary Dental Education and Research
Other Study IDs: AIDER-1301-AR
Record Dates: First submitted 2013-11-07; First posted 2013-11-20 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Oral Squamous Cell Carcinoma; Oral Epithelial Dysplasia
Keywords: Squamous Cell Carcinoma of the Head and Neck; Methyl Green Pyronin Staining; AgNORs; Morphometry
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples Without DNA — Oral mucosal biopsy specimens of study participants will be collected.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Normal or Control group: Those subjects with normal oral epithelium will be included in this group.
- Study Group: Those subjects with oral squamous cell carcinoma will be included in this group.

SUMMARY:
Oral cancer represents the sixth most common cancer worldwide whilst in Pakistan it ranks the second most common cancer in either gender. Histologically, over 90% of oral cancer lesions are squamous cell carcinomas which are diagnosed on the basis of histopathological analysis. However, proliferation kinetics and nucleolar status are not clearly delineated by routine H&E examination; thus making use of various proliferation markers imperative for the purpose.

Nuclear organizer regions (AgNORs) are associated with proliferative activity and represents as a diagnostic aid in oral malignancies. Similarly, methyl green pyronin (MGP) stain has also been valuable as a complement in routine histopathological studies of several neoplastic entities.

Morphometric techniques offer an opportunity to quantify nuclear changes associated with malignancy and may provide an objective basis for grading the tumors. The present study is planned to analyze the morphometric parameters of the MGP stain in oral squamous cell carcinoma, and in their various histological grades, and to assess if the MGP staining parameters could give information on the aggressiveness of the malignant lesions of oral cavity.

Sections from thirty cases of squamous cell carcinoma along with thirty cases of normal oral mucosa will be evaluated for methyl green pyronin (MGP) and AgNOR staining. Morphometric analysis of various MGP staining and AgNOR parameters would be performed using micrometer. Statistical analysis of the results will be carried out using SPSS. Quantitative variables will be expressed as mean ± Standard Deviation. Frequencies and percentages will be given for qualitative variables.

It is hypothesized that oral squamous cell carcinoma will exhibit significantly higher MGP staining and AgNOR staining parameters than normal mucosa of the oral cavity.

DETAILED DESCRIPTION:
Oral cancer, a major global health problem holds the sixth position worldwide with a marked variation in its geographic distribution. It is ranked as the third most frequent cancer in the developing world after stomach and cervical cancers. Amongst oral cancers, oral squamous cell carcinoma accounts for over 90% of the cases.

Out of the developing counties, Indo-Pak subcontinent amounts to one third of the global oral cancer burden. Carcinoma of the oral cavity in Pakistan, one of the high-risk countries is the second most frequent cancer in either gender. With differential distribution among sub-populations, it represents 8.8% of all reported cancer cases. The most predominant risk factors include tobacco smoking, betel chewing and alcohol.

Screening and specific diagnostic tools are two innovative approaches for early detection of oral cancer. Conventional oral examination and clinical evaluation remains the foundation of screening approaches whereas surgical biopsy followed by histological analysis is attributed to be the gold standard for diagnosing malignant oral lesions. Furthermore, some adjunctive techniques may contribute to the diagnosis of oral cancer. Of these vital staining, DNA analysis, chemiluminescence, tissue fluorescence, light-based detection systems and biomarkers are now on the forefront.

Biomarkers have been valuable in revealing additional information about tumor pathology, including the inactivation of tumor suppressor genes, angiogenesis, apoptosis and cell proliferation. Aberrations in proliferation kinetics are the most imperative factor during tumor progression. Three main categories of cell proliferation markers include growth fraction markers like Ki67, cycle-specific markers like PCNA(Proliferating Cellular Nuclear Antigen), and cell cycle time markers like AgNOR. During malignancy, proliferation and protein synthesis is mainly controlled by the nucleus.

Nucleolar Organizer Regions (NORs) are loops of DNA on the short arms of acrocentric chromosomes that presumably are associated with cell proliferation. Some of the NOR associated proteins are argyrophilic and can be demonstrated as black dots by the silver staining technique and the structures thus demonstrated are known as AgNORs. The AgNOR quantitative parameters provide information about the velocity of cell proliferation during cell cycle. Neoplastic progression is affected more by the rate of cell proliferation, rather than the proliferative activity per se.

Although AgNOR staining and AgNOR quantification are valuable methods in histopathological evaluation of malignancies, certain limitations have also been associated with this technique. Such AgNOR associated shortcomings include nucleolar affinity for silver stain obscuring the individual AgNORs in cases of intense staining, overlapping of variable degree between high and low grade tumors, difficulty in discerning doublets or clusters by light microscopy, misinterpreted stain deposition as proliferative activity along with some technical problems of staining and fixation.

Methyl Green Pyronin (MGP) stain is a differential stain used for selective staining of DNA and RNA. Methyl green binds specifically to deoxyribonucleic acid (DNA), staining nuclei green, while pyronin is specific for ribonucleic acid (RNA), staining nucleoli red. Methyl green pyronin stain has also been used to distinguish between proliferating and dedifferentiated non-proliferating cell nuclei. Similarly to assess the degradation of DNA in thyroid follicular epithelial cells, this stain has also proven to be useful.

Morphometry has been a significant advancement in delineating sequence of events responsible for cancer progression. Variations in nuclear and cellular size and shape have greater implications in the assessment of neoplastic lesions. Methyl Green Pyronin (MGP) stain has been attracting attention in the recent times as it has been used to evaluate various nuclear morphometric parameters in breast neoplasms. By using methyl green-pyronin staining, not only the inadequacies associated with AgNOR staining can be lessened but also the morphometric parameters for evaluating changes in the nucleus and nucleolus during carcinogenesis can be accomplished.

So far AgNOR staining appears to be a useful diagnostic tool in oral squamous cell carcinoma for examination of nucleolar structure and variations in nucleolar activity. On the other hand, MGP staining has been used in assessing the cancerous lesions of breast and thyroid gland and recently has been extended to oral lesions. However, no studies have been undertaken yet to evaluate and compare the morphometric parameters using these two stains within normal oral epithelium and oral squamous cell carcinoma. Similarly, very few studies have been undertaken regarding application of methyl green pyronin stain in oral pathologies.

Hence the current study has been planned to evaluate the morphometric parameters among normal oral epithelium and oral squamous cell carcinoma using methyl green pyronin staining; moreover these findings will also be compared with those of AgNOR staining. In this current scenario, methyl green pyronin staining and morphometric analysis may go hand in hand to provide a better diagnosis and early detection of oral cancer.

ELIGIBILITY:
Inclusion Criteria:

* Specimens of normal epithelium from healthy adult individuals irrespective of age and without habits that predispose to oral cancer
* Cases of clinically and histologically confirmed primary oral squamous cell carcinoma based on WHO criteria

Exclusion Criteria:

* Subjects of oral squamous cell carcinoma with any treatment therapy other than surgical excision.
* Subjects having metastatic tumors and tumors other than in the oral cavity
* Subjects having recurrent tumors.
* Subjects of normal or control group with history of risk / predisposing factors for oral cancer.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study population comprises of subjects reporting to dental departments of tertiary care hospitals of Lahore district in Pakistan.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Mean values of diameter, area and number of nuclei and nucleoli. | Within one week of staining of slides
  Morphometric parameters including diameter,area and number of nuclei and nucleoli will be determined using AgNOR and Methyl Green Pyronin staining methods.

SECONDARY OUTCOMES:
Association of grading of OSCC in relation to morphometric parameters | Within two weeks of staining of slides
  Chi-square test or Fisher exact test will be applied to see any statistical association of grading of OSCC in relation to morphometric parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Eyyaz Khaleel, M.Phil, Study Director — Postgraduate Medical Institute, Lahore; Ali Raza, B.D.S, Principal Investigator — Postgraduate Medical Institute, Lahore
Locations (1):
- Post Graduate Medical Institute, Lahore, Punjab Province, Pakistan

REFERENCES:
- [Background] Mohtasham N, Mahdavi-Shahri N, Salehinejad J, Ejtehadi H, Torabi-Parizi M, Ghazi N. Detection of nucleoproteins in squamous cell carcinoma, and dysplastic and normal mucosa in the oral cavity by methyl green-pyronin staining. J Oral Sci. 2010 Jun;52(2):239-43. doi: 10.2334/josnusd.52.239. PMID 20587947